CLINICAL TRIAL: NCT02710981
Title: Effect of Sildenafil Vaginal Gel Co-treatment With Clomiphene Citrate on Endometrial Thickness in Infertile Women With Prior Clomiphene Citrate Failure Due to Thin Endometrium: a Prospective Self-controlled Clinical Trial
Brief Title: Sildenafil Vaginal Gel Co-treatment With Clomiphene Citrate in Infertile Women With Thin Endometrium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Essam Rashad Abdel-Hafeez Othman, Associate professor, Assiut University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AUH1
Record Dates: First submitted 2016-03-04; First posted 2016-03-17 (Estimated); Results first posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Anovulation
Keywords: Sildenafil vaginal gel; endometrium; clomiphene; anovulation
MeSH Terms: conditions — Anovulation | interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clomiphene citrate only (Active Comparator): women with prior 5 ovulatory cycles of Clomiphene citrate induction, but without conception (clomiphene citrate failure), with thin endometrium (<8mm) in at least 3 cycles.
  Interventions: Drug: clomiphene citrate
- Sildenafil vaginal gel and Clomiphene (Experimental): Women who did not conceive on the Clomiphene citrate only cycle (41 women) were given Clomiphene citrate 100 mg/ day starting from day of the cycle for 5 days, with the addition to sildenafil vaginal gel 5 gm twice daily starting from day 8 of the cycle until day of HCG injection.
  Interventions: Drug: clomiphene citrate; Drug: Sildenafil vaginal gel

INTERVENTIONS:
Drug: clomiphene citrate — Clomiphene citrate only arm: Patients received Clomiphene citrate induction ( (in a dose of 100 mg/ day in two divided doses starting from day 3 of the cycle for 5 days) for the 6th cycle. A gel base, without medicament (vehicle only), was applied vaginally in a dose of 5 gm twice per day, from cycle day 8 to the day of HCG injection. Sonographic assessment of endometrial thickness together with Uterine artery Doppler evaluation were done in the late proliferative phase ( Day of HCG injection).
  Other Names: clomid only
Drug: Sildenafil vaginal gel — In addition to clomiphene citrate treatment as the previous group, women in the second arm were prescribed sildenafil vaginal gel in a dose of 5 g gel applied vaginally twice daily from cycle day 8 to the day of HCG injection. The sildenafil vaginal gel consists of sildenafil acetate as a medicament loaded on an in situ gelling system based on two polymers: Pluronic p-127, and Hydroxy Ethyl Cellulose.The gel was prepared in collaboration with the department of pharmaceutics, faculty of Pharmacy, Assiut University. Sixty grams of gel were prepared in tubes and every patient was given 10 applicators like that used for administration of vaginal antimycotic creams to use them for applying the gel.
  Other Names: Viagra vaginal gel
  Arms: Sildenafil vaginal gel and Clomiphene

SUMMARY:
This is a prospective self controlled clinical trial. Women with clomiphene Citrate failure, and thin endometrium were recruited (N = 42). In their 6th (Clomiphene citrate only) cycle, women continued on Clomiphene citrate 100 mg/ day for 5 days, and had sonographic measurement of their endometrial thickness , and Doppler evaluation of their uterine arteries on the day of HCG administration. In 7th cycle, women (N = 36) were given usual dose of Clomiphene citrate supplemented with sildenafil vagina gel (5 gm, containing 50 mg sildenafil) twice daily from cycle day 8 till the day of HCG injection. Endometrial thickness and uterine artery Doppler were measured on the day of HCG administration.

DETAILED DESCRIPTION:
Study design:

This is a prospective self-controlled clinical trial.

Study subjects:

Investigators counseled and recruited 42 infertile women who had been diagnosed with anovulatory infertility, with normal baseline FSH, LH, and free testosterone levels, patent tubes on hysterosalpingography, and normal male semen analysis.

By the time they were enrolled in the study, all women had already completed 5 ovulatory cycles of Clomiphene citrate induction (in a dose of 100 mg/ day in two divided doses starting from day 3 of the cycle for 5 days) but without conception (clomiphene citrate failure) with thin endometrium (<8mm) in at least 3 cycles. Ovulation was documented sonographically, and with day-21 serum progesterone exceeding 5 ng/ ml in all cases.

Exclusion criteria:

Women with major medical problems, male factor infertility, endocrine abnormalities such as hyperprolactinemia or abnormal thyroid functions, prior ovarian or adnexal surgery, or organic pelvic pathology were not included in the study.

Intervention:

Sixth cycle (Clomiphene citrate only):

Enrolled cases were asked to continue with Clomiphene citrate induction ( at the same dose) for the 6th cycle. A gel base, without medicament (vehicle only), was applied vaginally in a dose of 5 gm twice per day, from cycle day 8 to the day of HCG administration ( when follicular diameter reached 18 mm). Endometrial thickness and Uterine artery Doppler assessment were done in the late proliferative phase ( Day of HCG injection).

Seventh cycle ( Sildenafil vaginal gel and Clomiphene cycle):

Those who didn't conceive on the sixth cycle (41 women) were asked to have an extra (7th) cycle in which they were prescribed the usual dose of Clomiphene citrate in addition to sildenafil vaginal gel. The sildenafil vaginal gel consists of sildenafil acetate as a medicament loaded on an in situ gelling system based on two polymers: Pluronic p-127, and Hydroxy Ethyl Cellulose. The dose was 5 g gel containing 50 mg sildenafil, applied vaginally twice daily from cycle day 8 to Day of HCG injection. The gel was prepared in collaboration with the department of pharmaceutics, faculty of Pharmacy, Assiut University. Sixty grams of gel were prepared in tubes and every patient was given 10 applicators like that used for administration of vaginal antimycotic creams to use them for applying the gel.

Evaluation of the study end points:

On day of HCG injection (main follicular diameter of 18 mm) in the 6th, and 7th cycles, women came for follow up and had transvaginal sonographic assessment of their endometrial thickness. Investigators have measured the maximal distance spanning endometrial- myometrial interphase on each endometrial stripe in a sagittal plane in the fundus of the uterus. In addition, Transvaginal Doppler examination was also done on the same visit to evaluate the pulsatility indices of both uterine arteries. When the leading follicle reached 18 mm in diameter, 5000 IU of HCG was prescribed for IM injection.

Although pregnancy rate was not a primary outcome measure in the study, investigators detected pregnancy in 3 cases in the cohort of 36 cases of infertile women with clomiphene failure in which sildenafil gel was added as an adjuvant. Pregnancy was diagnosed with a B-HCG value above 100 mIU/ml, and confirmed later with ultrasound.

Statistics:

Data were analyzed using SPSS program ver. 17 using Student-t-test and Fisher's exact test for comparing data in the 6th and 7th cycles, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Women with clomiphene citrate failure (defined as at least prior 5 ovulatory cycles with clomiphene citrate, with no conception),
* persistently thin endometrium (less than 8 mm in at least 3 cycles).
* normal baseline FSH, LH, and free testosterone levels, patent tubes on hysterosalpingography, and normal male semen analysis

Exclusion Criteria:

* Women with major medical problems,
* male factor infertility,
* endocrine abnormalities such as hyperprolactinemia or abnormal thyroid functions,
* prior ovarian or adnexal surgery, or organic pelvic pathology

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed N. Fetih, M.D., Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As this is a self controlled clinical trial, participants in the clomiphene citrate only arm (6th ovulation induction cycle) are the same participant in the clomiphene citrate plus sildenafil vaginal gel arm (7th ovulation induction cycle).
Groups:
- Clomiphene Citrate Only: Clomiphene citrate only arm: Patients underwent 6th ovulation induction cycle in which women received Clomiphene citrate (in a dose of 100 mg/ day in two divided doses starting from day 3 of the cycle for 5 days). A gel base, without medicament (vehicle only), was applied vaginally in a dose of 5 gm twice per day, from cycle day 8 to the day of HCG injection. Sonographic assessment of endometrial thickness together with Uterine artery Doppler evaluation were done in the late proliferative phase ( Day of HCG injection). Period of this arm is one menstrual cycle (6th induction cycle)
- Clomiphene Citrate Plus Sildenafil Vaginal Gel (7th Ovulation): Clomiphene citrate plus sildenafil vaginal gel arm: Women who did not conceive on the 6th cycle ( clomiphene citrate only cycle; 41 women) were offered a 7th cycle in which they were given Clomiphene citrate 100 mg/ day starting from day of the cycle for 5 days, with adding sildenafil vaginal gel 5 gm twice daily starting from cycle day 8 on until day of HCG injection. Sonographic assessment of endometrial thickness together with Uterine artery Doppler evaluation were done in the late proliferative phase ( Day of HCG injection). Period of this arm is the subsequent menstrual cycle (7th induction cycle)
Period: 6th Ovulation Induction Cycle (5 Days)
Arm/Group | Clomiphene Citrate Only | Clomiphene Citrate Plus Sildenafil Vaginal Gel (7th Ovulation)
Started | 42 | 0
Completed | 41 | 0
Not Completed | 1 | 0
Period: 7th Ovulation Induction Cycle (5 Days)
Arm/Group | Clomiphene Citrate Only | Clomiphene Citrate Plus Sildenafil Vaginal Gel (7th Ovulation)
Started | 0 | 41
Completed | 0 | 36
Not Completed | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Clomiphene Citrate Only Group (6th Ovulation Induction Cycle): Infertile women who have completed 5 cycles of clomiphene citrate with successful ovulation, thin endometrium and no pregnancy who are attempting a 6th cycle of clomiphene citrate.
Arm/Group | Clomiphene Citrate Only Group (6th Ovulation Induction Cycle)
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 41
Serum FSH [Mean (Standard Deviation); unit: U/L] | 4.5 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Endometrial Thickness
Description: Transvaginal sonographic measurement of maximal distance spanning endometrial- myometrial interphase on each endometrial stripe in a sagittal plane in the fundus of the uterus
Time Frame: Day of HCG administration
Measure: Mean (Standard Deviation); unit: millimeter
Groups:
- Clomiphene Citrate Only Group (6th Ovulation Induction Cycle): Infertile women who had undergone 5 cycles of clomiphene citrate ovulation induction with ovulation detected, and no pregnancy due to thin endometrium
- Clomiphene Citrate Plus Sildenafil Vaginal Gel (7th Ovulation): Women who did not get pregnant after 6th ovulation induction cycle receive a 7th induction cycle with clomiphene citrate plus sildenafil vaginal gel
Arm/Group | Clomiphene Citrate Only Group (6th Ovulation Induction Cycle) | Clomiphene Citrate Plus Sildenafil Vaginal Gel (7th Ovulation)
Number analyzed (Participants) | 41 | 36
millimeter | 6.6 (1.4) | 9.3 (3.1)

2. Secondary Outcome: Uterine Blood Flow
Description: Doppler ultrasound is used to measure the pulsatility index in both uterine arteries. Pulsatility index is a measure of the arterial resistance to blood flow. The higher the value of the pulsatility index, the more resistant the uterine arteries are, and hence the worst the outcome.
Time Frame: Day of HCG administration
Measure: Mean (Standard Deviation); unit: index
Groups:
- Clomiphene Citrate Plus Sildenafil Vaginal Gel (7th Ovulation): Women who did not get pregnant after 6th ovulation induction cycle with clomiphene citrate and placebo vaginal gel were offered a 7th cycle in which ovulation was induced with clomiphene citrate plus sildenafil vaginal gel
Arm/Group | Clomiphene Citrate Only Group (6th Ovulation Induction Cycle) | Clomiphene Citrate Plus Sildenafil Vaginal Gel (7th Ovulation)
Number analyzed (Participants) | 41 | 36
index | 2.4 (0.8) | 1.6 (1.3)

3. Secondary Outcome: Clinical Pregnancy Rate
Description: Identifying pregnancy through positive urinary HCG test plus sonographic detection of cardiac pulsations
Time Frame: At the end of a 28-day menstrual cycle.
Measure: Count of Participants; unit: Participants
Groups:
- Clomiphene Citrate Plus Sildenafil Vaginal Gel (7th Ovulation: Women who did not get pregnant after 6th ovulation induction cycle with clomiphene citrate and placebo vaginal gel were offered a 7th ovulation induction cycle with clomiphene citrate and sildenafil vaginal gel
Arm/Group | Clomiphene Citrate Only Group (6th Ovulation Induction Cycle) | Clomiphene Citrate Plus Sildenafil Vaginal Gel (7th Ovulation
Number analyzed (Participants) | 41 | 36
Participants | 0 | 3

ADVERSE EVENTS:
Groups:
- Clomiphene Citrate Only Group (6th Ovulation Induction Cycle): Infertile women who had undergone 5 cycles of clomiphene citrate ovulation induction with ovulation detected, and no pregnancy due to thin endometrium (N =41)
Arm/Group | Clomiphene Citrate Only Group (6th Ovulation Induction Cycle) | Clomiphene Citrate Plus Sildenafil Vaginal Gel (7th Ovulation)
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clomiphene Citrate Only Group (6th Ovulation Induction Cycle) (N=41) | Clomiphene Citrate Plus Sildenafil Vaginal Gel (7th Ovulation) (N=36)
Vasodilatory headache (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No